CLINICAL TRIAL: NCT06918327
Title: The Power of Concentrated Growth Factor: A New Era in Pain Management in Third Molar Surgery
Brief Title: Effect of CGF on Postoperative Pain After Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mert Zeytinoğlu, Assoc. Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGE-DHF-MZ-002
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Oral Complication
Keywords: Pain; Third molar; VAS scale
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGF (Experimental): Participants received CGF after the operation on one side
  Interventions: Other: Concentrated Growth Factor; Other: non-CGF
- non-CGF (No Intervention): The other extraction socket is left empty

INTERVENTIONS:
Other: Concentrated Growth Factor — Bilaterally impacted third molar of the patients are removed surgically and concentrated growth factor is placed in one of the extraction sockets.
  Arms: CGF
Other: non-CGF — The other extraction socket is left empty for control purposes.
  Arms: CGF

SUMMARY:
The purpose of this study is to evaluate the effects of concentrated growth factor (CGF) on pain after bilateral impacted third molar surgery and to determine its contribution to the healing process.

The main question it aims to answer is:

Is CGF effective on reducing the pain in impacted third molar surgery? Researchers compare the pain on the CGF-applied and CGF free sides after impacted third molar surgery. Postoperative pain is assessed using the Visual Analogue Scale. TThe postoperative outcomes including pain are clinically assessed at different-time intervals (1-7 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral, symmetrical, bone-retained (vertical, mesioangular, horizontal) impacted wisdom teeth in the mandible, regardless of gender
* Patients without any systemic disease
* Patients who have been informed about the duration, purpose and requirements of the study and who have signed the informed consent form voluntarily.

Exclusion Criteria:

* Having a disease affecting general health that requires the application of prophylactic antimicrobial agents
* Having a systemic viral, fungal or bacterial infection
* Patients with acute or chronic maxillary sinusitis
* Suspected or diagnosed pregnancy and nursing mothers
* Patients with heart and vascular diseases
* Patients with liver disease, haematological disease and neoplastic disease
* Patients who have recently received anti-inflammatory therapy
* Patients with chronic medication use (antihistamines, NSAIDs, steroids and antidepressants)
* Patients predisposed to psychotic or psychopathic tendencies
* Patients with rheumatic diseases, blood diseases, diabetes mellitus
* Patients at cardiological risk of infective endocarditis
* Patients under antibiotic pressure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain on CGF-applied and CGF free sides in bilateral impacted third molar surgery | The postoperative outcomes including pain are clinically assessed at different-time intervals (1st, 2nd, 3rd, 4th, 5th, 6th and 7th days).
  The primary outcome measure is postoperative pain on CGF-applied and CGF free sides in bilateral impacted third molar surgery. Postoperative pain is assessed using the Visual Analogue Scale (VAS). Patients are asked to mark the pain they felt on the scale (10 cm long line) on the (1-7) days after the operation. The end of the line indicates unbearable pain, the beginning indicates no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Zeytinoğlu, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No